CLINICAL TRIAL: NCT02910219
Title: Diarrhea Prevention and Prophylaxis With Crofelemer in HER2 Positive Breast Cancer Patients Receiving Trastuzumab, Pertuzumab, and Docetaxel or Paclitaxel With or Without Carboplatin: HALT-D
Brief Title: Diarrhea Prevention and Prophylaxis With Crofelemer in HER2 Positive Breast Cancer Patients
Acronym: HALT-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sandra Swain (Other)
Collaborators: Lombardi Comprehensive Cancer Center (Other); Medstar Health Research Institute (Other); Genentech, Inc. (Industry); Napo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Sandra Swain, Medical Oncologist, Georgetown University
Organization: Georgetown University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MHRI GU 2015-0547
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Results first posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: HER2; pertuzumab; trastuzumab; docetaxel; paclitaxel; carboplatin; crofelemer; chemotherapy induced diarrhea
MeSH Terms: conditions — Breast Neoplasms | interventions — crofelemer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crofelemer (Experimental): Patients on the treatment arm will take one tablet of crofelemer twice a day (each tablet is 125 mg), to be swallowed whole without chewing or crushing, during cycles 1-2 of chemotherapy with THP or TCHP. Patient will be monitored off crofelemer during cycle 3 of chemotherapy.
  Interventions: Drug: Crofelemer
- Control (No Intervention): Patients on the control arm will be on the study for cycles 1-3 of THP or TCHP. Patients on the control arm will not receive crofelemer at any time on this study.

INTERVENTIONS:
Drug: Crofelemer — Crofelemer 125 mg BID during cycles 1-2 of THP or TCHP
  Arms: Crofelemer

SUMMARY:
Chemotherapy induced diarrhea is seen in up to 40-80% of patients receiving this treatment for HER2 positive locally advanced or metastatic breast cancer. This diarrhea can significantly impact a patient's quality of life and ability to tolerate chemo/anti-HER2 therapy. This study will look at the efficacy of the drug crofelemer in preventing diarrhea in breast cancer patients.

DETAILED DESCRIPTION:
Various anti-diarrheal agents, such as loperamide, codeine, octreotide, are available for diarrhea management, but few are used in the prophylactic setting and none provide a targeted approach for treating chemotherapy induced diarrhea (CID).

Pre-clinical studies have suggested that blocking EGFR results in excess chloride secretion and thus diarrhea. Crofelemer is an extract from the blood red bark of Croton lechleri that inhibits luminal chloride efflux by blocking the calcium activated chloride channel (CaCC) and cystic fibrosis transmembrane regulator (CFTR) chloride channels. Due to its size and polarity, it acts only luminally and is not systemically absorbed. It is currently FDA approved for use in preventing diarrhea in HIV/AIDS patients on anti-retroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent;
2. Men and women ≥18 years of age;
3. Pathologically confirmed diagnosis of HER2 positive breast cancer of any stage (previous treatment is allowed without limits on lines of prior therapy);
4. Scheduled to receive at least 3 consecutive cycles of THP or TCHP;
5. Performance status of 0-2 according to the ECOG scale;
6. Negative pregnancy test at time of informed consent for women of childbearing potential;
7. Able to read, understand, follow the study procedure and complete crofelemer, rescue medication, and bowel movement diaries;
8. Patients may enroll simultaneously on this study and other studies, including but not limited to NSABP B52;
9. Patients with brain metastases (including concurrent steroid treatment) are allowed on this study.
10. Left Ventricular Ejection Fraction (LVEF) greater or equal to 50% at baseline as determined by either ECHO or MUGA

Exclusion Criteria:

1. Pregnant and/or breastfeeding;
2. Ongoing irritable bowel syndrome (IBS) or colitis (including but not limited to ulcerative colitis, Crohn's disease, microscopic colitis, etc.);
3. Use of investigational drugs within 3 weeks of signing consent or foreseen use during the study;
4. Use of chemotherapy, trastuzumab, or pertuzumab within the past 3 weeks;
5. Use of antibiotics within the past 7 days (up to 2 prophylactic doses of antibiotics for procedures including, but not limited to port placement, is permitted);
6. Any type of ostomy;
7. Total colectomy;
8. Fecal incontinence;
9. Ongoing radiation induced diarrhea or constipation or planned radiotherapy to the abdomen or pelvis while on study;
10. Active systemic infection requiring ongoing intervention, including but not limited to oral and intravenous antibiotics, anti-fungals, anti-parasites, anti-virals;
11. Abdominal or pelvic surgery without recovery of bowel function;
12. Inadequate organ function for starting THP or TCHP, which may include the following laboratory results within 28 days prior to signing consent:

    1. Total bilirubin > upper limit of normal (ULN) (unless the patient has documented Gilbert's syndrome)
    2. Serum creatinine > 2.0 mg/dL or 177 μmol/L
    3. AST (SGOT) and ALT (SPGT) > 2.5 ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - MedStar Franklin Square Cancer Center at Loch Raven Campus, Baltimore, Maryland
  - Harry and Jeanette Weinberg Cancer Institute, Baltimore, Maryland
  - John Theurer Cancer Center at Hackensack Univ, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data available

REFERENCES:
- [Background] Gao JJ, Tan M, Pohlmann PR, Swain SM. HALT-D: A Phase II Evaluation of Crofelemer for the Prevention and Prophylaxis of Diarrhea in Patients With Breast Cancer on Pertuzumab-Based Regimens. Clin Breast Cancer. 2017 Feb;17(1):76-78. doi: 10.1016/j.clbc.2016.08.005. Epub 2016 Aug 27. PMID 27692565
- [Derived] Pohlmann PR, Graham D, Wu T, Ottaviano Y, Mohebtash M, Kurian S, McNamara D, Lynce F, Warren R, Dilawari A, Rao S, Mainor C, Swanson N, Tan M, Isaacs C, Swain SM. HALT-D: a randomized open-label phase II study of crofelemer for the prevention of chemotherapy-induced diarrhea in patients with HER2-positive breast cancer receiving trastuzumab, pertuzumab, and a taxane. Breast Cancer Res Treat. 2022 Dec;196(3):571-581. doi: 10.1007/s10549-022-06743-9. Epub 2022 Oct 25. PMID 36280642

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Crofelemer | Control
Started | 27 | 26
Completed | 26 | 25
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Patients on the treatment arm will take one tablet of crofelemer twice a day (each tablet is 125 mg), to be swallowed whole without chewing or crushing, during cycles 1-2 of chemotherapy with THP or TCHP. Patient will be monitored off crofelemer during cycle 3 of chemotherapy.
  Crofelemer: Crofelemer 125 mg BID during cycles 1-2 of THP or TCHP
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Full Range); unit: years] | 53.9 [27 to 78.5] | 52 [27 to 78.5] | 52.9 [27 to 78.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 14 | 17 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Diarrhea for >= 2 Consecutive Days
Description: Percentage of participants with any grade (based on CTCAE 4.0) diarrhea lasting 2 or more consecutive days during cycles 1 and 2 of chemotherapy.
Time Frame: Cycle 1, Cycle 2 (each cycle is 21 days)
Measure: Number; unit: percentage of patients
Arm/Group | Crofelemer | Control
Number analyzed (Participants) | 26 | 25
percentage of patients
  Cycle 1 | 68 | 69.6
  Cycle 2 | 65.2 | 72.2

2. Secondary Outcome: Diarrhea Any Grade
Description: Incidence of diarrhea of any grade, as measured by CTCAE v4.0, by cycle
Time Frame: Cycle 1, Cycle 2 (each cycle is 21 days)
Population: The number analyzed is different from overall number due to early treatment discontinuation.
Measure: Count of Participants; unit: Participants
Arm/Group | Crofelemer | Control
Number analyzed (Participants) | 26 | 25
Participants
  Cycle 1 (investigator-assessed) | 16 | 16
  Cycle 2 (investigator-assessed): number analyzed (Participants) | 25 | 23
  Cycle 2 (investigator-assessed) | 15 | 18

3. Secondary Outcome: Grade 3-4 Diarrhea
Description: number of patients with diarrhea of grade 3 or grade 4, as measured by CTCAE v4.0, by cycle and by stratum
Time Frame: Cycle 1, Cycle 2 (each cycle is 21 days)
Population: The number analyzed is different from overall number due to early treatment discontinuation.
Measure: Count of Participants; unit: Participants
Arm/Group | Crofelemer | Control
Number analyzed (Participants) | 26 | 25
Participants
  Cycle 1 | 1 | 2
  Cycle 2: number analyzed (Participants) | 25 | 23
  Cycle 2 | 0 | 4

4. Secondary Outcome: Diarrhea Onset
Description: Time to onset of first episode of diarrhea of any grade, overall
Time Frame: from baseline through Cycle 3 (21 day cycles)
Population: The number analyzed is different from overall number due to missing data.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Crofelemer | Control
Number analyzed (Participants) | 25 | 23
days | 3 [1 to 4] | 2 [1 to 4]

5. Secondary Outcome: Diarrhea Duration
Description: Duration (days) of any grade diarrhea, defined from day 1 to day 21, by cycle in which the episode started
Time Frame: Cycle 1, Cycle 2 (each cycle is 21 days)
Population: Duration of the "FIRST day of diarrhea" to the "LAST day of diarrhea" based on patient diary. Only Cycle 1 and Cycle 2 analyzed. The number analyzed is different from overall number due to missing data.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Crofelemer | Control
Number analyzed (Participants) | 25 | 23
days
  Cycle 1 | 13 [8 to NA] — NA = upper confidence limit of infinity | 15 [10 to NA] — NA = upper confidence limit of infinity
  Cycle 2: number analyzed (Participants) | 23 | 18
  Cycle 2 | 15 [9 to NA] — NA = upper confidence limit of infinity | 12 [9 to NA] — NA = upper confidence limit of infinity

6. Secondary Outcome: Duration Grade 3-4 Diarrhea
Description: Duration (days) of grade 3-4 diarrhea during cycle 1 through the end of cycle 2, defined from cycle day 1 to cycle 2 day 21
Time Frame: End of Cycle 2 (each cycle is 21 days)
Measure: Mean (Full Range); unit: days
Arm/Group | Crofelemer | Control
Number analyzed (Participants) | 1 | 4
days | 18 [0 to 18] | 6.5 [1 to 12]

7. Secondary Outcome: Anti-diarrheal Medications
Description: Use of anti-diarrheal medications (other than study drug), by cycle and arm
Time Frame: Cycle 1, Cycle 2 (each cycle is 21 days)
Population: Only cycle 1 and cycle 2 analyzed. Total amount of Loperamide, Diphenoxylate Atropine and Octreotide; No subjects in the Crofelemer arm received octreotide in either cycle 1 or 2.
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Crofelemer | Control
Number analyzed (Participants) | 26 | 22
units
  Cycle 1- Loperamide | 20.69 (36.74) | 24.73 (41.4)
  Cycle 2-Loperamide: number analyzed (Participants) | 24 | 22
  Cycle 2-Loperamide | 16.25 (23.43) | 21.24 (31.52)
  Cycle 1-Diphenoxylate Atropine | 16.15 (82.36) | 2.272 (12.79)
  Cycle 2- Diophnoxylate Atropine: number analyzed (Participants) | 24 | 21
  Cycle 2- Diophnoxylate Atropine | 0.8333 (3.18) | 5.595 (25.64)
  Cycle 1- Octreotide | 0 (0) | 6.818 (31.98)
  Cycle 2- Octreotide: number analyzed (Participants) | 24 | 21
  Cycle 2- Octreotide | 0 (0) | 71.43 (327.3)

8. Secondary Outcome: FACIT-D Total Score
Description: Quantitative FACIT-D (FACIT-D Functional Assessment of Chronic Illness Therapy for Patients With Diarrhea) total score, collected day 1 of each cycle and at the time of study completion, cycles 1 and 2 reported; The higher the score the better the QOL; Score range 0-152.
Time Frame: Cycle 1, Cycle 2 (each cycle is 21 days)
Population: The number analyzed is different from overall number due to early treatment discontinuation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crofelemer | Control
Number analyzed (Participants) | 26 | 25
score on a scale
  Cycle 1 | 129.0 (14.3) | 123.8 (20.4)
  Cycle 2: number analyzed (Participants) | 25 | 23
  Cycle 2 | 116.7 (19.8) | 114.4 (23.3)

9. Secondary Outcome: FACIT-D Diarrhea Score
Description: Quantitative FACIT-D (FACIT-D Functional Assessment of Chronic Illness Therapy for Patients With Diarrhea) diarrhea subscale (DS) score, by cycle; Score Range 0-44; the higher the score, the better the QOL.
Time Frame: Cycle 1, Cycle 2 (each cycle is 21 days)
Population: The number analyzed is different from overall number due to early treatment discontinuation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crofelemer | Control
Number analyzed (Participants) | 26 | 25
score on a scale
  Cycle 1 | 40.5 (6.2) | 39.8 (6.3)
  Cycle 2: number analyzed (Participants) | 25 | 23
  Cycle 2 | 34.9 (6.8) | 34.1 (7.8)

10. Secondary Outcome: Stool Frequency Based on Consistency (Bristol Stool Scale)
Description: Frequency of stool consistency of 6-7, as measured by the Bristol Stool scale (minimum 1-separate hard lumps, maximum 7-watery, no solid pieces), by cycle; Median in watery bowel movements (Bristol Stool Form Scale 6-7).
Time Frame: Cycle 1, Cycle 2 (each cycle is 21 days)
Population: The number analyzed is different from overall number due to early treatment discontinuation.
Measure: Median (Full Range); unit: number of bowel movements
Arm/Group | Crofelemer | Control
Number analyzed (Participants) | 26 | 25
number of bowel movements
  Cycle 1: number analyzed (Participants) | 25 | 23
  Cycle 1 | 14.5 [0 to 102] | 19 [4 to 72]
  Cycle 2: number analyzed (Participants) | 23 | 18
  Cycle 2 | 14.0 [0 to 139] | 17.5 [1 to 75]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from signing consent to 30 days after completing study or 30 days after last dose of crofelemer, whichever occurs later (until cycle 4 day 1).
Arm/Group | Crofelemer | Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/26 | 7/25
Other Adverse Events (participants affected / at risk) | 26/26 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crofelemer (N=26) | Control (N=25)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) — port-a-cath infection
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1) — Cellulitis
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crofelemer (N=26) | Control (N=25)
Anemia (Blood and lymphatic system disorders) | 5 (8) | 3 (5)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 18 (116) | 22 (93)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 10 (12) | 12 (15)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 10 (12) | 9 (10)
Infusion related reaction (General disorders) | 0 (0) | 3 (3)
Pain (General disorders) | 3 (4) | 3 (3)
Alanine aminotransferase increased (Investigations) | 2 (6) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (4) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (6) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Dysgeusia (Nervous system disorders) | 3 (5) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 4 (5)
Anxiety (Psychiatric disorders) | 4 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3)
Weight loss (Investigations) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT02910219/Prot_SAP_000.pdf